CLINICAL TRIAL: NCT06906952
Title: A Prospective Single-center Randomized Controlled Trial of Robotic Surgery With Transrectal Resection Specimens (NOSES-IV) and Traditional Assisted Robotic Surgery for the Treatment of High Rectal and Sigmoid Colon Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchang University (Other)
Responsible Party: Principal Investigator, Taiyuan Li, professor, Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZL078
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Natural Orifice Specimen Extraction Surgery; Robotic Surgery; Short-term Outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOSES-IV Group (Experimental): After the body is free, the tumor segment of the bowel is pulled out through the anus. Excise the tumor segment of the colon outside the anus.
  Interventions: Procedure: robotic natural orifice specimen extraction surgery
- non-NOSES Group (Sham Comparator): After internal mobilization, the tumor segment of the bowel was removed through an abdominal incision. Excise the tumor segment of the bowel outside the incision.
  Interventions: Procedure: robotic transabdominal specimen extraction surgery

INTERVENTIONS:
Procedure: robotic natural orifice specimen extraction surgery — After the rectum and its mesorectum were dissociated, the rectum was transected at 2 cm below the tumor by using a linear stapler. Then the rectal stump was incised and disinfected with iodophor, the protective sleeve was placed into the abdominal cavity through the assistant hole. An assistant delivered oval forceps into the pelvic cavity through the anus and used oval forceps to grip one end of the protective sleeve. Then slowly pulled out the protective sleeve. Eventually, one end of the protective sleeve was placed inside the abdominal cavity and the other outside the anus, completely covering the rectal stump and the perianal area. Tumor was pulled out of the rectal stump, then the colon was then disconnected at 10 cm above the tumor. The anvil was placed into the stump of the sigmoid colon and disinfected with iodophor, and then the anvil was delivered into the abdominal cavity. Place a circular stapler through the anus for end-to-end anastomosis of the rectum and sigmoid colon.
  Arms: NOSES-IV Group
Procedure: robotic transabdominal specimen extraction surgery — After the rectum and its mesorectum were dissociated, the rectum was transected at 2 cm below the tumor by using a linear stapler. Take a 6cm incision through the rectus abdominis muscle in the lower left abdomen and place an incision protective cover. Cut off the intestinal tube 10cm from the upper edge of the tumor and place a stapler base. The rectal stump was sutured with purse-string suture. Place a circular stapler through the anus for end-to-end anastomosis of the rectum and sigmoid colon. After completion of digestive tract reconstruction. The pelvic and abdominal cavities were washed repeatedly with normal saline until there were no blood remained. Close the abdominal cavity layer by layer.
  Arms: non-NOSES Group

SUMMARY:
This study aimed to compare the short-term efficacy of robotic radical resection of high rectal cancer and sigmoid colon cancer (NOSES-IV) with transrectal resection specimens and traditional robotic surgery in the treatment of high rectal cancer and sigmoid colon cancer. At the same time, the safety and advantages of robotic radical resection of high rectal cancer and sigmoid colon cancer (NOSES-IV) with transrectal resection specimens and traditional robotic surgery in the treatment of high rectal cancer and sigmoid colon cancer were compared.

ELIGIBILITY:
Inclusion Criteria:

* 1) The age is more than 18 years old and less than or equal to 85 years old 2) Eastern Cooperative Oncology Group score ≤2 3) Preoperative pathological diagnosis of rectal adenocarcinoma 4) cT1-3NxM0 rectal cancer defined by preoperative contrast-enhanced MRI 5) The maximum diameter of tumor ≤5cm on preoperative enhanced MRI 6) The body can tolerate the operation and sign the informed consent

Exclusion Criteria:

* 1) multiple primary colorectal cancer 2) recurrent rectal cancer 3) preoperative neoadjuvant chemoradiotherapy 4) complicated with intestinal obstruction or intestinal bleeding requiring emergency surgery 5) previous anal surgery history 6) BMI≥30kg/m2 7) severe mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The rate of all complications | 1 months after surgery
  incidence rate
The rate of all complications (Clavien-Dindo grade ≥ III ) | 1 months after surgery
  incidence rate

SECONDARY OUTCOMES:
operative time | Intraoperative
  minutes
estimation of blood loss | Intraoperative
  milliliters
postoperative hospital stay | 1 day after operation
  days
visual analogue pain score | 1 weeks after surgery
  score

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi 330000, Nanchang, China

IPD SHARING:
Plan to Share IPD: No